CLINICAL TRIAL: NCT01554488
Title: Inhaled Fluticasone Effects on Upper Airway Patency in Obstructive Lung Disease
Acronym: InFLOW
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low subject accrual
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLIN-20-11S
Record Dates: First submitted 2012-02-29; First posted 2012-03-15 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea
Keywords: asthma; COPD; sleep apnea, obstructive
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): High dose inhaled fluticasone (1760mcg/day)
  Interventions: Drug: Inhaled Fluticasone Propionate
- Arm 2 (Active Comparator): Low dose inhaled fluticasone (88mcg/day)
  Interventions: Drug: Inhaled Fluticasone Propionate

INTERVENTIONS:
Drug: Inhaled Fluticasone Propionate — Inhaled corticosteroid

SUMMARY:
The Chairman of the Veterans' Disability Benefits Commission reported at a recent US Senate hearing that asthma, chronic obstructive pulmonary disease (COPD), and sleep apnea are among the top 13 most frequent diagnoses leading to disability under the Department of Defense and the VA system statutes. Recent research finds that sleep apnea is more common among asthma and COPD individuals, and this may be caused by inhaled corticosteroid use. Many Veterans are currently using inhaled corticosteroids, and many more will be prescribed such medications, given their recent inclusion in international treatment guidelines. As such, this study addresses a critical need by researching the role of a potent inhaled corticosteroid in promoting sleep apnea, the determinants of this response, and the ways through which it occurs. Results from this study will form the foundation for future research aimed at expanding understanding of the effects of inhaled corticosteroids on the upper airway, as well as developing means to prevent or counteract them.

DETAILED DESCRIPTION:
BACKGROUND: Growing data suggest that patients with obstructive lung disease (OLD) such as asthma and chronic obstructive pulmonary disease (COPD) have an increased predisposition for obstructive sleep apnea, but the mechanism(s) remain unknown. One characteristic these patients share is use of inhaled corticosteroid (ICS). The investigators recently found a dose-dependent relationship of ICS use with high OSA risk. Furthermore, in a 16-week observational inhaled fluticasone (FP) treatment study, the investigators observed increased upper airway (UAW) collapsibility during sleep, as measured by the critical closing pressure (Pcrit), paralleling the improvement in lower airways obstruction, with the largest Pcrit deterioration in the subject with most sleep-disordered breathing (SDB) at baseline. These findings suggest an effect of ICS on the "unified airway" of steroid responsive patients and of those with more collapsible upper airways at baseline. The investigators also found a dose-dependent relationship of ICS with obesity. Based on their known effects, ICSs could deleteriously affect UAW collapsibility through inducing dilators' myopathy and fat deposition around the UAW. FP is the most potent and commonly used ICS.

HYPOTHESIS/AIMS: The central hypothesis is that FP will increase UAW collapsibility (less negative Pcrit) and worsen SDB in steroid responsive patients with OLD and those with UAWs more susceptible to collapse at baseline, through alterations in tongue muscle function and fat accumulation in the UAW surrounding structures. To address this hypothesis, the investigators propose to test the effects of inhaled FP on: 1) UAW collapsibility during sleep and SDB severity, assessed by Pcrit, measured as we previously reported (1) and polysomnographic (PSG) measures. Exploratory aims will test the role of steroid responsiveness and baseline collapsibility as determinants of FP effects on Pcrit and SDB; 2) tongue strength and fatigability, and fat accumulation (fraction and volume, measured on MRI) in the surrounding UAW structures, measured as we previously reported (1,2).

DESIGN: The investigators propose a proof-of-concept and mechanistic, randomized-controlled, parallel groups study of high (220 mcg, 4 puffs twice a day) vs. low (44 mcg twice a day) dose inhaled FP, followed by an 8-week wash-out period, in 58 steroid-naive subjects with OLD. Following baseline Pcrit, PSG, MRI and tongue function, subjects will enter a 2-week low-dose FP run-in, with subsequent randomization to either high- vs. low-dose FP, for 16 weeks. At mid-period, Pcrit, tongue function and steroid responsiveness status (defined as 5% improvement from baseline in FEV1%) will be determined. At the end of treatment, Pcrit, PSG, MRI and tongue measurements will be taken. Then, subjects will enter an 8-week wash-out that ends with repeat Pcrit and tongue function assessments.

SIGNIFICANCE: Millions of people, including many Veterans, are treated with ICS for OLD, and among those with COPD, these numbers are likely to escalate. However, do these medications alter UAW collapsibility and predispose to OSA in some individuals, as the investigators' preliminary observations suggest? This research is innovative because it will directly evaluate the effects of ICS on the UAW structure and function during sleep and wakefulness. At the study completion, it is the investigators expectation that they will have elucidated the effects and governing mechanisms of ICS on UAW patency and SDB severity. Data generated will form the foundation for future research aimed at expanding the investigators' understanding of ICS's effects on UAW and means to mitigate/prevent them. The clinical implication of these findings will be experimental-based verification of deleterious effects of ICS on UAW and risk for OSA, which will ultimately be of enormous financial benefit to the VA and OLD management programs.

ELIGIBILITY:
Inclusion Criteria:

* American Veterans
* age 18 and above
* diagnosis of asthma and COPD per guidelines
* for asthma, persistent symptoms per guidelines
* for asthma, a pre-bronchodilator FEV1 55-90% and DLCO 80% predicted
* for asthma, physiologic confirmation by bronchodilator or methacholine challenge
* for COPD, a post-bronchodilator ratio of FEV1/FVC 70% and FEV1 50%
* overall smoking history of <10 pack-years for asthma and 10 pack-years for COPD.

Exclusion Criteria:

* any use of inhaled corticosteroid for >2 weeks at a time during the last 6 months, or any use in the last 6 weeks;
* as needed use of nasal steroids in the prior 6 months
* select medications
* recent exacerbation requiring oral or systemic steroids in the past 6 months
* diagnosed vocal cords dysfunction
* other lung diseases (lung cancer, sarcoidosis, tuberculosis, lung fibrosis) or known 1-antitrypsin deficiency
* significant or actively unstable medical or psychiatric illnesses
* diagnosed osteopenia or osteoporosis
* established diagnosis of neuromuscular disease
* BMI 45 kg/m2 and higher
* treated OSA
* pregnancy (confirmed on urine test) or desire to get pregnant in the upcoming 6 months.
* smoking in the past 6 months
* metallic or electronic implants
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Teodorescu, MD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

REFERENCES:
- [Background] Teodorescu M, Xie A, Sorkness CA, Robbins J, Reeder S, Gong Y, Fedie JE, Sexton A, Miller B, Huard T, Hind J, Bioty N, Peterson E, Kunselman SJ, Chinchilli VM, Soler X, Ramsdell J, Loredo J, Israel E, Eckert DJ, Malhotra A. Effects of inhaled fluticasone on upper airway during sleep and wakefulness in asthma: a pilot study. J Clin Sleep Med. 2014 Feb 15;10(2):183-93. doi: 10.5664/jcsm.3450. PMID 24533002
- [Background] Humbert IA, Reeder SB, Porcaro EJ, Kays SA, Brittain JH, Robbins J. Simultaneous estimation of tongue volume and fat fraction using IDEAL-FSE. J Magn Reson Imaging. 2008 Aug;28(2):504-8. doi: 10.1002/jmri.21431. PMID 18666214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects enrolled 3/12/2013-11/6/2015
Pre-assignment Details: 28 subjects were eligible at V2 and entered the 2-week low dose fluticasone run-in phase, necessary to assess fluticasone adherence. Thereafter, three subjects withdrew consent and were not randomized. Thus, 25 subjects were randomized.
Groups:
- High Dose Inhaled Fluticasone: High dose inhaled fluticasone (1,760mcg/day)
- Low Dose Inhaled Fluticasone: Low dose inhaled fluticasone (88mcg/day)
  Inhaled Fluticasone Propionate: Inhaled corticosteroid
Period: Overall Study
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Started | 13 | 12
Completed | 12 | 9
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- High Dose Inhaled Fluticasone: High dose inhaled fluticasone (1760mcg/day)
  Inhaled Fluticasone Propionate: Inhaled corticosteroid
- Total: Total of all reporting groups
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (18) | 37.3 (14) | 42.2 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 5 | 14
Asthma [Count of Participants; unit: Participants] — Population: The subject population also included those with COPD for which the numbers are reported in the next section.
  Participants
    randomized | 9 | 11 | 20
    completed the study: number analyzed (Participants) | 12 | 9 | 21
    completed the study | 8 | 8 | 16
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] — Population: subject population included those with asthma, reported in the previous section
  Participants
    randomized | 4 | 1 | 5
    completed the study: number analyzed (Participants) | 12 | 9 | 21
    completed the study | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Upper Airway Critical Closing Pressure (Pcrit) at Week 16
Description: Pressure at which the pharyngeal upper airway closes during stable non-REM sleep, measured as described in the referenced citation.
Time Frame: 16-week randomized controlled phase
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 12 | 9
cmH2O | -3.03 (3.66) | -1.68 (2.16)
Statistical Analysis 1: Comparison: High Dose Inhaled Fluticasone vs Low Dose Inhaled Fluticasone; All of the comparisons were based on mixed effects linear regression models with visit and group*visit as fixed effects and subject as a random effect. Confidence intervals for the treatment difference (group*visit interaction) were constructed using the Wald method; Test type: Other; Mean Difference (Net) = -1.03, 95% CI 2-sided [-5.03 to 2.92]

2. Secondary Outcome: Tongue Strength at Anterior Location at Week 16
Description: Wakefulness tongue function was measured using the Iowa Oral Performance Instrument (IOPI) at anterior and posterior tongue locations, as described in the referenced citation. In brief, this instrument has a small-sized, air-filled plastic balloon, called sensor or bulb, which was inserted between the tongue blade and the roof of the mouth. At each location, the tongue strength was determined as the maximum pressure generated against the IOPI bulb during a forced tongue contraction. Several standardized trials were conducted to ensure reproducibility.
Time Frame: 16-week randomized phase
Measure: Mean (Standard Deviation); unit: KiloPascals
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 12 | 9
KiloPascals | 61 (14.4) | 63.7 (18.5)

3. Secondary Outcome: Tongue Strength at Posterior Location at Week 16
Description: as for outcome 2
Time Frame: 16-week randomized phase
Measure: Mean (Standard Deviation); unit: KiloPascals
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 12 | 9
KiloPascals | 55.5 (11.7) | 58.1 (16.7)

4. Secondary Outcome: Tongue Fatigability at Anterior Location at Week 16
Description: Wakefulness tongue function was measured using the Iowa Oral Performance Instrument (IOPI) at anterior and posterior tongue locations, as described in the referenced citation. In brief, this instrument has a small-sized, air-filled plastic balloon, called sensor or bulb, which was inserted between the tongue blade and the roof of the mouth. At each location, the tongue strength was determined as the maximum pressure generated against the IOPI bulb during a forced tongue contraction. Then, tongue fatigability was measured through a submaximal task, as the time (in seconds) able to maintain > 50% of the above measured strength, at each location. Several standardized trials were conducted for each measure and at each location, to ensure reproducibility.
Time Frame: 16-week randomized treatment phase
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 12 | 9
seconds | 74.4 (53.3) | 78 (25.5)

5. Secondary Outcome: Tongue Fatigability of Posterior Location at Week 16
Description: as for outcome 4
Time Frame: 16-week randomized treatment phase
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 12 | 9
seconds | 53 (18) | 65.9 (23.7)

6. Other Pre Specified Outcome: Tongue Volume at Week 16
Description: Tongue volume was assessed on Magnetic Resonance (MR) imaging of the area extending from the level of the roof of the hard palate to the vocal cords, with the subject awake and lying on their back. We used a specialized technique called Iterative Decomposition of water and fat with Echo Asymmetry and Least squares estimation Fast Spin-Echo (IDEAL-FSE), developed at University of Wisconsin by our collaborator and used for assessing the tongue (2). In brief, at first, the method provides well co-registered, separate water and fat images, which are free from the artifact that corrupts the usual MR images. Subsequently, these separate images are recombined in new high resolution images which provide: 1) comprehensive anatomical reference to delineate the tongue and measure its volume, and; 2) unambiguous separation of adipose tissue, to allow determination of fat volume and fraction in the tongue.
Time Frame: 16-week randomized treatment phase
Population: 1 subject in High dose and 2 subjects in Low dose inhaled fluticasone groups had contraindications, eg, metal in their bodies (2) or claustrophobia (1) and could not undergo MRI testing, per the set exclusion criteria.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 11 | 7
mm^3 | 73.2 (15.5) | 75.9 (15)

7. Other Pre Specified Outcome: Percentage Fat Content (Fat Fraction) of the Tongue at Week 16
Description: Tongue fat content was assessed on Magnetic Resonance (MR) imaging of the area extending from the level of the roof of the hard palate to the vocal cords, with the subject awake and lying on their back. We used a specialized technique called Iterative Decomposition of water and fat with Echo Asymmetry and Least squares estimation Fast Spin-Echo (IDEAL-FSE), developed at University of Wisconsin by our collaborator and used for assessing the tongue (2). In brief, at first, the method provides well co-registered, separate water and fat images, which are free from the artifact that corrupts the usual MR images. Subsequently, these separate images are recombined in new high resolution images which provide: 1) comprehensive anatomical reference to delineate the tongue and measure its volume, and; 2) unambiguous separation of adipose tissue, to allow determination of fat volume and fraction in the tongue.
Time Frame: 16-week randomized controlled phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of total tongue volume
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 11 | 7
percentage of total tongue volume | 27.8 (9.98) | 24.6 (7.88)

8. Other Pre Specified Outcome: Volume of Pharyngeal Upper Airway Surrounding Structures at Week 16
Description: The volume of pharyngeal upper airway surrounding structures was assessed on Magnetic Resonance (MR) imaging, as we published (1). We scanned the area extending from the level of the roof of the hard palate to the vocal cords, with the subject awake and lying on their back, We used a specialized technique called Iterative Decomposition of water and fat with Echo Asymmetry and Least squares estimation Fast Spin-Echo (IDEAL-FSE). In brief, at first, the method provides well co-registered, separate water and fat images, which are free from the artifact that corrupts the usual MR images. Subsequently, these separate images are recombined in new high resolution images which provide: 1) comprehensive anatomical reference to delineate the tongue and measure its volume, and; 2) unambiguous separation of adipose tissue, to allow determination of fat volume and fraction in the upper airway structures.
Time Frame: 16-week randomized controlled phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 11 | 7
mm^3 | 205 (67.9) | 194 (73.7)

9. Other Pre Specified Outcome: Percentage Fat Content (Fat Fraction) of Pharyngeal Upper Airway Surrounding Structures at Week 16
Description: Pharyngeal upper airway fat content was assessed on Magnetic Resonance (MR) imaging, as we published (1). We scanned the area extending from the level of the roof of the hard palate to the vocal cords, with the subject awake and lying on their back, We used a specialized technique called Iterative Decomposition of water and fat with Echo Asymmetry and Least squares estimation Fast Spin-Echo (IDEAL-FSE). In brief, at first, the method provides well co-registered, separate water and fat images, which are free from the artifact that corrupts the usual MR images. Subsequently, these separate images are recombined in new high resolution images which provide: 1) comprehensive anatomical reference to delineate the tongue and measure its volume, and; 2) unambiguous separation of adipose tissue, to allow determination of fat volume and fraction in the upper airway structures.
Time Frame: 16-week randomized controlled phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of total airway volume
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Number analyzed (Participants) | 11 | 7
percentage of total airway volume | 41.5 (24.6) | 31.5 (17.4)

ADVERSE EVENTS:
Time Frame: from study initiation up to 16 weeks of randomized treatment. In addition, monitoring continued for an additional two months step-down inhaled fluticasone treatment under medical supervision by the study team.
Arm/Group | High Dose Inhaled Fluticasone | Low Dose Inhaled Fluticasone
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/9
Other Adverse Events (participants affected / at risk) | 6/12 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Inhaled Fluticasone (N=12) | Low Dose Inhaled Fluticasone (N=9)
needed gallbladder surgery for stones (Hepatobiliary disorders) | 1 (1) | 1 (1) — subject with chronic obstructive pulmonary disease (COPD) developed acute cholecystitis due to stones, had endoscopic retrograde cholangio-pancreatography, and ultimately needed cholecystectomy.
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — subject with asthma, in the low fluticasone dose group, developed an exacerbation requiring prednisone bursts
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Inhaled Fluticasone (N=12) | Low Dose Inhaled Fluticasone (N=9)
tongue lesion from broken tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
broken tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
yeast infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early due to low accrual. The original scientific question remains unanswered. Based on the experience with this study, a multi-center study would be necessary to accrue sufficient participants to answer the question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes